CLINICAL TRIAL: NCT00681473
Title: Late Effects of Proton Radiation Therapy in Patients With Low-Grade Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-195
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Low Grade Gliomas
Keywords: proton radiation therapy; photon radiation therapy
MeSH Terms: interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiation Therapy (Experimental): Proton radiation therapy daily (Monday through Friday) for six weeks. This is a single arm study.
  Interventions: Radiation: Proton Radiation Therapy

INTERVENTIONS:
Radiation: Proton Radiation Therapy — Once daily, Monday through Friday, for 6 weeks.

SUMMARY:
In this research study, we are looking to study the side effects from the use of proton radiation in treating people with low-grade gliomas that are recommended radiation treatment. We expect response of the tumors to be the same with proton radiation as compared to standard 3D conformal radiation therapy, but also expect less side effects from radiation.

DETAILED DESCRIPTION:
* Participants will receive radiation therapy for 6 weeks, given in daily doses, Monday through Friday, for a total of 30 treatments.
* A medical history and physical examination will be performed prior to the start of radiation treatment, weekly during the 6 weeks of radiation and after the finish of radiation performed at 3 and 6 months and then annually for 5 years.
* Hormonal function tests will be taken prior to the start of radiation treatment and after the finish of radiation treatment at 3 and 6 months, and annually for five years to assess the participants hormonal functions as they relate to the pituitary gland's function.
* A brain MRI will be performed prior to the start of radiation treatment and then performed at 3 and 6 months after radiation treatment then annually for 5 years.
* A neurocognitive exam will be performed prior to the start of radiation therapy, a limited exam 6 months after the completion of radiation therapy, and a complete exam annually for 5 years.
* Quality of Life and Emotional Well-Being Questionnaires will be done before radiation begins, 2 months after radiation treatment, 6 months after radiation treatment and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed low-grade gliomas, WHO classification II/IV or equivalent low grade histology, including protoplasmic, fibrillary, gemistocytic astrocytomas, and mixed variants such as oligoastrocytomas
* Must have at least one of: (1) progressive or recurrent disease as defined by imaging, (2) persistence or progression of debilitating neurological symptoms, or (3) at risk of early progression as defined by either (a) age of 40 or older or (b) MIB-1 of 3% or greater
* KPS of 70 or greater
* 18 years of age or older
* Surgical and medical/chemotherapeutic interventions are per physician's discretion and are acceptable
* Must be able to speak and comprehend English

Exclusion Criteria:

* Other baseline neurocognitive or emotional disorders or deficits, including but not limited to head injury, CVA, TIA, or other cerebral insults with residual neuropsychiatric deficits, psychiatric disorders, learning disabilities, HIV positivity or other medical conditions at high risk of causing neurocognitive decline or emotional instability
* Prior history of cranial irradiation
* Pregnancy at the time of radiation treatment
* Unable to undergo MRI scans (e.g., embedded ferromagnetic metal or pacemakers)
* Comorbid illness or reason to suggest a life expectancy of less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen A. Shih, MD, MS, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A large number of patients with brain tumors in the greater area are referred to one or more of the MGH multidisciplinary brain tumor specialists for evaluation and further care.
Period: Overall Study
Arm/Group | Proton Radiation Therapy
Started | 20 (20 patients with WHO Grade 2 Glioma were enrolled.)
Completed | 20 (All 20 patients completed RT and tolerated treatment well.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 20 baseline participants were included in analysis.
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 37.5 [22 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Late Effects > 3 Months Post RT
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Percentage of Participants With Progression Free Survival
Description: Clinical and/or radiographic assessments Percentages were estimated by Kaplan Meier
Time Frame: At 1, 3, and 5 years
Measure: Number; unit: % of participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 20
% of participants
  1 Year | 100
  3 Year | 85
  5 Year | 40

3. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Percentages were estimated by Kaplan Meier
Time Frame: At 1, 3, and 5 years
Measure: Number; unit: % of participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 20
% of participants
  1 Year | 100
  3 Year | 95
  5 Year | 84

ADVERSE EVENTS:
Time Frame: Up to 5 years post RT
Arm/Group | Proton Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation Therapy (N=20)
fatigue, acute (General disorders) | 20 (20)
Erythema (Skin and subcutaneous tissue disorders) | 17 (17)
Headache, acute (General disorders) | 15 (15)
Seizure, acute (Nervous system disorders) | 5 (5)
Taste/Smell Alteration, acute (General disorders) | 3 (3)
Anorexia (General disorders) | 2 (2)
Alopecia, acute (Skin and subcutaneous tissue disorders) | 17 (17)
Cognitive Deficit (Nervous system disorders) | 1 (1)
Nausea/Vomiting, acute (Gastrointestinal disorders) | 4 (4)
Paresthesia, acute (General disorders) | 2 (2)
Dizziness, acute (Nervous system disorders) | 2 (2)
Anxiety (Nervous system disorders) | 2 (2)
Insomnia, acute (General disorders) | 2 (2)
Motor Dysfunction (Nervous system disorders) | 2 (2)
Photophobia (Eye disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Hearing (Ear and labyrinth disorders) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Temperature Sensitivity (General disorders) | 3 (3)
Weakness, cranial nerve (Nervous system disorders) | 3 (3)
Weakness, peripheral (Nervous system disorders) | 2 (2)
Stuttering, twitching (General disorders) | 1 (1)
Cognitive dysarthria (Nervous system disorders) | 1 (1)
Visual disturbance, other than loss (Eye disorders) | 3 (3)
Vision Loss (Eye disorders) | 1 (1)
Proprioceptive deficit (Nervous system disorders) | 1 (1)
fatigue, late (General disorders) | 17 (17)
headache, late (Gastrointestinal disorders) | 15 (15)
Seizure, late (Nervous system disorders) | 4 (4)
Taste/smell alteration, late (General disorders) | 1 (1)
Alopecia, late (Skin and subcutaneous tissue disorders) | 12 (12)
Nausea/Vomiting, late (Gastrointestinal disorders) | 3 (3)
Paresthesia, late (General disorders) | 3 (3)
Dizziness, late (Nervous system disorders) | 6 (6)
Insomnia, late (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes